CLINICAL TRIAL: NCT06854237
Title: Prevalence and Characteristics of Widespread Pain in People With Knee Osteoarthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: KOA WSP 284125
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Widespread Chronic Pain
Keywords: Knee osteoarthritis; Widespread pain; Pain sites; Correlation
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis: Patients with knee osteoarthritis will perform the 30 seconds chair stand test to evaluate physical performance and compare with self-reported pain history and number of pain locations.

SUMMARY:
The goal is to evaluate whether the number of pain sites or pain estimation with Instant and Constant Osteoarthritis Pain (ICOAP) is related to functional impairment in the lower extremity in people with knee osteoarthritis (KOA).

The main questions it aims to answer are:

1. What is the relationship between the number of pain sites and physical function when adjusted for age, sex, education level, and origin in people with KOA?
2. What is the relationship between pain experience measured with ICOAP (constant and intermittent pain subscales, as well as total score) and reduced physical function when adjusted for age, sex, education level, and origin in people with KOA?
3. What is the relationship between demographic data (age, sex, BMI, origin, level of education) and reduced physical function in people with KOA?

Participants were recruited from five rehabilitation clinics in primary care within the Västra Götaland region, for another study (NCT03855813). Patients with diagnosed KOA were asked to participate in the study. The patients mostly had problems in the knee joint but could also have osteoarthritis (OA) in other joints.

DETAILED DESCRIPTION:
Background

Knee osteoarthritis (KOA) affects approximately 14% of the Swedish population over the age of 45 (1). Typical symptoms are pain, stiffness and reduced physical function (2). Most people with KOA (90%) have at least two pain sites (3). One-third of people with chronic knee pain meet criteria for widespread pain, which is associated with impaired self-rated physical function (4, 5). Female gender, ethnic background, synovitis and degree of osteoarthritis (OA) on X-ray are predictors of a deterioration in function in people with OA in the lower extremity (6). Multiple pain sites are associated with fear of movement (3), while increased fear of movement has a moderate correlation with reduced physical function in people with KOA (7). While high self-efficacy can predict an increased physical function (7).

Evaluating leg muscle strength can be critical in identifying people with OA who are at risk of worsening and who may need to strengthen their muscles to improve physical function and relieve pain. This may also help prevent sarcopenia and its metabolic consequences (8). Today, self-assessment forms and performance-based tests are used to assess patients' physical function (9). An advantage of performance-based tests compared to self-assessment forms is that they measure what the patient is actually able to do (10), and performance-based tests are better at differentiating between pain and physical function (11). These tests are usually performed in the clinic under the supervision of healthcare personnel.

For people who do not have the ability to perform functional testing, pain history can be of value in differentiating whether or not a person has lower extremity functional limitations - without being evaluated with tests or forms. Because pain in people with OA can vary, assessment with the ICOAP form can be used to describe whether the pain changes (12). However, lack of time can prevent clinics from using standardized forms or instruments (13).

More knowledge is needed that describes how common it is with widespread pain among people with KOA who seek primary care and examine the relationship between pain intensity, number of pain sites, and its impact on function, activity and quality of life. In addition, it is of interest to examine relationships between demographic data and pain history on physical function in order to assess the functional impairment according to a standardized function test with the help of common anamnesis questions in the clinical meeting with the patient without having to perform the actual test. The knowledge of these correlations is missing today.

Purpose

The aim of this study is to evaluate whether the number of pain sites or pain estimation with ICOAP is related to a functional impairment in the lower extremity in people with KOA.

Research questions:

1. What is the relationship between the number of pain sites and physical function when adjusted for age, sex, education level and origin for people with KOA?
2. What is the relationship between pain experience measured with ICOAP (constant and intermittent pain subscales, as well as total score) and reduced physical function when adjusted for age, sex, education level and origin of people with KOA?
3. What is the relationship between demographic data (age, sex, BMI, origin, level of education) and reduced physical function for people with KOA?

Method: Population/Sample

Inclusion criteria

Participants were recruited from five rehab clinics in primary care within the Västra Götaland region to a former study which this study is based on (NCT03855813). Patients with diagnosed KOA were asked to participate in the study. The patients mostly had problems in the knee joint, but could also have OA in other joints in the lower extremities. They were independent in walking, with or without walking aids, and could understand test instructions both verbally and in writing in Swedish.

Exclusion criteria

* Neurological problems that affected balance or walking ability.
* Severe or serious somatic or mental illnesses that affected the ability to function or the ability to understand and follow the test instructions.
* Had knee or hip replacement in the past six months.
* Other knee surgery in the last six months that could affect functional capacity.

Method: Data collection

Patients with established KOA received written information about the study, consent form and questionnaire about background data, either directly at the clinic or by written letter. When participating in the study, the patients filled in all the forms at home and brought them to the physiotherapist at the next visit.

Background data

Background data included age, sex, body mass index (BMI), other diseases, pain sites, pain intensity, duration of pain in the knee joint and experience of the knee problems.

Pain history

Pain intensity was measured with a numeric rating scale (NRS) 0-10 (14), where 0 corresponds to no pain and 10 the worst imaginable pain. The patient rated the pain at rest, when loaded, and on average over the past week.

ICOAP - the Swedish version, was used to assess the pain experience. The questionnaire contains two subscales with question areas about intermittent and constant pain. The total score for the subscale for intermittent pain varies between 0-24 points and between 0-20 points for constant pain. The total score, 0-44 points, is usually recalculated to a scale of 0-100 (total score/44 x 100), where 0 corresponds to no pain and 100 to extreme pain (12).

The number of pain sites was evaluated with a pain drawing with 18 predefined body areas (15).

Functional test with 30 CST

The chair test "30 seconds chair stand test" (30 CST) is part of a test battery that is recommended both in research and in the clinic for people with OA. This test is a reliable and valid method for measuring the strength and functional capacity of people with OA assessed by clinician (16, 17), and as a self-test (18).

The chair test 30 CST was performed on an approximately 45 cm high chair without armrests. The participant was asked to do as many stands as possible in 30 seconds. The starting position was sitting on the chair. The stands would be to an upright position (fully extended hips and knees), then back to a seated position. The arms were to be crossed over the chest throughout the test. In all measurements with the chair test, the patient had to indicate perceived pain intensity in the knee joint before and during the test. All physiotherapists received training on the study protocol and the chair test.

Method: Data processing/Data analysis

Sample size

The sample size was calculated with the statistical program PASS 16, for the reliability study for which the data for this study is based on (18). Sample size of 117 participants, with two observations per participant for each inter- and intra-rater test, achieved a power of 80% to detect an intraclass correlation coefficient (ICC) of 0.8 with a significance level of 0.05. A total of 114 participants were recruited for the reliability study. All participants in the reliability study (n=114) will be included in this study and are considered to be sufficiently plentiful to be able to answer the purpose and the research questions with good probability.

Statistical analysis

Demographic data will be presented in the form of central and dispersion measures depending on the data level. For nominal data, number and percent are presented.

Logistic regression will be conducted between the independent variables 1) demographic data, 2) number of pain sites, 3) ICOAP to assess the effects on the dependent variable impaired physical function measured by 30 CST. The results from the regression analysis will be presented with the odds ratio with 95% confidence interval and illustrated with graphs of the expected probabilities. The analyzes will be carried out in the statistical program Statistical Package for Social Science (SPSS) (19). The significance level is set at p< 0.05.

Expected meaning

The number of pain sites could be used to detect potential risks in functional impairment and could be helpful to clinicians when deciding how to treat patients with KOA, without having to spend time on functional tests. This patient group with multiple pain sites may need more support to maintain physical activity. An understanding of possible effects between people's background history and physical function could contribute to people with KOA being able to receive more individually tailored and preventive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed knee osteoarthritis, could have problems/osteoarthritis in other joints, but the knee joint should have been the most troublesome.
* Independent in walking, with och without walking aids.
* Understand test instructions both verbally and in writing in Swedish.

Exclusion Criteria:

* Neurological problems that affected balance or walking ability.
* Severe or serious somatic or mental illnesses that affected the ability to function or the ability to understand and follow the test instructions.
* Completed knee or hip replacement in the past six months.
* Other knee surgery in the past six months that could affect physical functional capacity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed knee osteoarthritis, with or without problems/osteoarthritis in other joints, but the knee joint should have been the most troublesome.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical function | One occasion at baseline
  Measured with 30 seconds chair stand test. The participant is asked to stand up from a chair as many times as possible during 30 seconds. A higher number of stands indicate a better physical function.
Osteoarthritis pain | One occasion at baseline
  Osteoarthritis pain will be measured with Measure of Intermittent and Constant Osteoarthritis Pain: ICOAP. The questionnaire consists of two subscales, a) constant pain and b) intermittent pain. The total score ranges between 0 to 100 where 0 means no pain and 100 means extreme pain.
Pain locations | One occasion at baseline
  Self-reporting pain assessment with pre-defines locations on a pain drawing.

SECONDARY OUTCOMES:
Pain intensity | One occasion at baseline
  Pain intensity was measured with a numeric rating scale (NRS) 0-10 (14) , where 0 corresponds to no pain and 10 the worst imaginable pain. The patient rated the pain at rest, when loaded, and on average over the past week.

OTHER OUTCOMES:
Demographic data | Baseline
  Demographic data such as age, sex, body mass index (BMI), duration osteoarthritis diagnosis, other diseases, education level, origin, pain duration (knee). Patients' body weight and height will be measured to calculate the BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Mei Ho-Henriksson, MD, Principal Investigator — Västra Götalandsregionen, Närhälsan, Närhälsan Lidköping Rehabmottagning, Lidköping, Sweden
Locations (1):
- Närhälsan Lidköping Rehabmottagning, Lidköping, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to General Data Protection Regulation, to protect the participant's privacy.

REFERENCES:
- [Background] Gill S, Hely R, Page RS, Hely A, Harrison B, Landers S. Thirty second chair stand test: Test-retest reliability, agreement and minimum detectable change in people with early-stage knee osteoarthritis. Physiother Res Int. 2022 Jul;27(3):e1957. doi: 10.1002/pri.1957. Epub 2022 May 19. PMID 35592902
- [Background] Gill S, McBurney H. Reliability of performance-based measures in people awaiting joint replacement surgery of the hip or knee. Physiother Res Int. 2008 Sep;13(3):141-52. doi: 10.1002/pri.411. PMID 18697226
- [Background] Bergman S, Herrstrom P, Hogstrom K, Petersson IF, Svensson B, Jacobsson LT. Chronic musculoskeletal pain, prevalence rates, and sociodemographic associations in a Swedish population study. J Rheumatol. 2001 Jun;28(6):1369-77. PMID 11409133
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Turner GM, Litchfield I, Finnikin S, Aiyegbusi OL, Calvert M. General practitioners' views on use of patient reported outcome measures in primary care: a cross-sectional survey and qualitative study. BMC Fam Pract. 2020 Jan 24;21(1):14. doi: 10.1186/s12875-019-1077-6. PMID 31980021
- [Background] Hawker GA, Davis AM, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Katz JN, Dieppe P. Development and preliminary psychometric testing of a new OA pain measure--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):409-14. doi: 10.1016/j.joca.2007.12.015. PMID 18381179
- [Background] Stratford PW, Kennedy DM, Woodhouse LJ. Performance measures provide assessments of pain and function in people with advanced osteoarthritis of the hip or knee. Phys Ther. 2006 Nov;86(11):1489-96. doi: 10.2522/ptj.20060002. PMID 17079748
- [Background] Terwee CB, Mokkink LB, Steultjens MP, Dekker J. Performance-based methods for measuring the physical function of patients with osteoarthritis of the hip or knee: a systematic review of measurement properties. Rheumatology (Oxford). 2006 Jul;45(7):890-902. doi: 10.1093/rheumatology/kei267. Epub 2006 Feb 3. PMID 16461441
- [Background] Jordan KP, Wilkie R, Muller S, Myers H, Nicholls E; Arthritis Research Campaign National Primary Care Centre. Measurement of change in function and disability in osteoarthritis: current approaches and future challenges. Curr Opin Rheumatol. 2009 Sep;21(5):525-30. doi: 10.1097/BOR.0b013e32832e45fc. PMID 19525848
- [Background] Sanada K, Iemitsu M, Murakami H, Gando Y, Kawano H, Kawakami R, Tabata I, Miyachi M. Adverse effects of coexistence of sarcopenia and metabolic syndrome in Japanese women. Eur J Clin Nutr. 2012 Oct;66(10):1093-8. doi: 10.1038/ejcn.2012.43. Epub 2012 May 9. PMID 22569087
- [Background] Odole A, Ekediegwu E, Ekechukwu END, Uchenwoke C. Correlates and predictors of pain intensity and physical function among individuals with chronic knee osteoarthritis in Nigeria. Musculoskelet Sci Pract. 2019 Feb;39:150-156. doi: 10.1016/j.msksp.2018.11.014. Epub 2018 Nov 28. PMID 30623891
- [Background] Sandhar S, Smith TO, Toor K, Howe F, Sofat N. Risk factors for pain and functional impairment in people with knee and hip osteoarthritis: a systematic review and meta-analysis. BMJ Open. 2020 Aug 7;10(8):e038720. doi: 10.1136/bmjopen-2020-038720. PMID 32771991
- [Background] Aydemir B, Muhammad LN, Song J, Chang AH, Dunlop DD, Chang RW, Lee YC. Modifiable physical and behavioural factors associated with widespread pain in older adults with radiographic evidence of knee osteoarthritis. Musculoskeletal Care. 2023 Dec;21(4):1090-1097. doi: 10.1002/msc.1789. Epub 2023 Jun 4. PMID 37271894
- [Background] Turkiewicz A, Petersson IF, Bjork J, Hawker G, Dahlberg LE, Lohmander LS, Englund M. Current and future impact of osteoarthritis on health care: a population-based study with projections to year 2032. Osteoarthritis Cartilage. 2014 Nov;22(11):1826-32. doi: 10.1016/j.joca.2014.07.015. Epub 2014 Jul 30. PMID 25084132
- [Background] Peral Perez J, Mortensen SR, Lluch Girbes E, Gronne DT, Thorlund JB, Roos EM, Skou ST. Association between widespread pain and psychosocial factors in people with knee osteoarthritis: a cross-sectional study of patients from primary care in Denmark. Physiother Theory Pract. 2025 Apr;41(4):752-762. doi: 10.1080/09593985.2024.2372381. Epub 2024 Jul 1. PMID 38946473
- [Background] Bergman S, Thorstensson C, Andersson MLE. Chronic widespread pain and its associations with quality of life and function at a 20- year follow-up of individuals with chronic knee pain at inclusion. BMC Musculoskelet Disord. 2019 Dec 9;20(1):592. doi: 10.1186/s12891-019-2976-3. PMID 31818282
- See also: Research database, Research and development in Region Västra Götaland — https://www.researchweb.org/is/se/vgr/project/284125